CLINICAL TRIAL: NCT04426630
Title: An Accessible, Scalable, Patient-facing mHealth Application for Self-care of Heart Failure in LMIC
Brief Title: mHealth for Self-care of Heart Failure in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Makerere University (Other); Uganda Heart Institute (Other); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000025338; 1R21TW010998-01A1 (NIH)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Results first posted 2022-08-10 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure
Keywords: Heart Failure; Telemedicine; Uganda; mHealth; Implementation Science
MeSH Terms: conditions — Heart Failure | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: This is a single-center prospective cohort study. The researchers will use consecutive sampling to identify potential patient participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mHealth (Other): Heart failure patients enrolled in the mHealth program
  Interventions: Other: mHealth for heart failure patients in Uganda

INTERVENTIONS:
Other: mHealth for heart failure patients in Uganda — Patients at Uganda Heart Institute will be enrolled in an mHealth program intended to promote self-care for heart failure and improve their healthcare quality of life.

SUMMARY:
Heart failure affects more than 38 million people globally. It is responsible for high rates of hospitalization and premature mortality, especially in sub-Saharan Africa. Heart failure causes multiple debilitating and distressing symptoms. These symptoms can often be managed by patients themselves but only when they are able to identify symptoms and select appropriate actions. Self-care, a World Health Organization-endorsed intervention for chronic conditions like heart failure, is greatly underutilized in lower and middle income countries, including Uganda. Self-care refers to the ability of patients, caregivers and communities to maintain health, prevent disease, and manage illness, with or without a healthcare provider. Mobile health (mHealth) offers a promising platform to address this need gap in lower and middle income countries. mHealth takes advantage of the widespread usage of mobile phones to offer patients individualized self-care tools such as education, healthy lifestyle prompts, and support with making decisions. Since 2016, this multidisciplinary, international research team has been designing Medly Uganda, an mHealth application to improve self-care among Ugandan patients with heart failure. This application began as a smartphone but was adapted for the low-cost feature phones used widely throughout the country. It was also integrated into an mHealth system endorsed by the Ugandan Ministry of Health. When patients log in they are prompted to report on specific heart failure symptoms. The application then generates self-care instructions based on those symptoms. If a patient reports serious symptoms the application triggers an alert to the research nurse, who then consults with the patient, caregiver, and if needed, cardiologist, to establish a plan of care. This study proposes that an mHealth intervention tailored specifically to the local context will improve healthcare quality of life for patients with heart failure. The research team hypothesizes that heart failure patients who use the program will report improved scores on the Self-Care in Heart Failure Index. These scores will be assessed at baseline, three-month, and six-month visits. The researchers will also measure changes in patients' clinical conditions, including the 6-minute walk test, left ventricular ejection fraction, and frequency of acute care visits. Finally, the researchers will conduct qualitative interviews with patients and providers to understand their experiences.

DETAILED DESCRIPTION:
Participants will be asked to initiate self-care sessions using the Medly Uganda application. They will dial the sub-code and enter a unique PIN to access the system. They are asked to do this every Monday, Wednesday, and Friday morning for six months, as well as anytime that they experience concerning symptoms. If a participant has not initiated a session by 11:00am on the designated days, the application will generate an SMS reminder. Each interactive session will present a series of symptom-based questions to the participant. These questions will be followed by a tailored SMS message. While session content will not remain on the participant's phone, the SMS messages will. This allows participants to retain and review messages, thereby reinforcing educational content. There are four status categories: Stable, Fluid Overload, Urgent, and Critical. If Stable, participants will be sent one of six encouraging and educational messages. If Fluid Overload, Urgent or Critical, patient participants will be sent a message that identifies the symptom and recommends an action and the on-duty nurse will be sent an accompanying alert. Urgent and Critical alerts will also be sent to the on-duty doctor. The nurse is expected to call the patient for Urgent and Critical alerts within 60 and 15 minutes, respectively. Nurse phone call interactions will be guided by a standard operating manual. One nurse and one doctor will be designated rotating 'on-duty' responsibility to monitor clinician alerts and the dashboard seven days a week. The doctor will be available to provide clinical supervision to the nurse as needed and they will have a daily in-person or by-phone.

ELIGIBILITY:
Inclusion Criteria:

* UHI patient presenting for routine or urgent outpatient visit
* Currently living in Uganda and not planning to travel abroad for six months
* Age >=18 years
* Symptomatic heart failure (New York Heart Association Class II or III and left ventricular ejection fraction of 45% or less)
* Access to a mobile phone
* Basic reading skills in English, Luganda, and/or Runyankole

Exclusion Criteria:

* Life expectancy < six months
* Active medical condition requiring hospitalization, such as cardiac ischemia (acute electrocardiographic changes and/or positive biomarkers, if available), syncope, or significant fluid overload
* Pregnancy
* Inability to provide informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Schwartz, MD, Principal Investigator — Yale University; Isaac Ssinabulya, MMed, Principal Investigator — Uganda Heart Institute
Locations (1):
- Uganda Heart Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- mHealth: Heart failure patients in Uganda were enrolled in an mHealth program at the Uganda Heart Institute. The program intended to promote self-care for heart failure and improve patient healthcare quality of life.
Period: Overall Study
Arm/Group | mHealth
Started | 72
Completed | 66
Not Completed | 6
Not completed — Death | 4
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | mHealth
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 2
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53.0 [40.0 to 65.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 72
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 72
Healthcare Quality of Life: EQ-5D [Count of Participants; unit: Participants] — Healthcare quality of life will be measured using the 5-level EQ-5D version (EQ-5D-5L). It is a validated instrument appropriate for use in lower and middle income countries. Each of the five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) comprises the EQ-5D descriptive system. We regrouped the 5 levels of perceived problems into binary responses as "no problem" (Level 1), or "Having problems" (Level 2-5).
  Participants
    Mobility: No Problem | 47
    Mobility: Having Problems | 25
    Self-Care: No Problem | 42
    Self-Care: Having Problems | 30
    Usual Activities: No Problem | 33
    Usual Activities: Having Problems | 39
    Pain or Discomfort: No Problem | 42
    Pain or Discomfort: Having Problems | 30
    Anxiety or Depression: No Problem | 44
    Anxiety or Depression: Having Problems | 28
Health Quality of Life: EQ VAS [Median (Inter-Quartile Range); unit: units on a scale] — The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the 100 indicates 'The best health you can imagine' and 0 means 'The worst health you can imagine'.
  units on a scale | 70 [50 to 80]

OUTCOME MEASURES:

1. Primary Outcome: Self-Care for Heart Failure Index, Maintenance
Description: The Self-care of Heart Failure Index (SCHFI) is a measure of self-care defined as a naturalistic decision-making process involving the choice of behaviors that maintain physiological stability (maintenance), the response to symptoms when they occur (management), and confidence in self-care (confidence). The self-care maintenance subscale includes 10 items asking how often patients check their heart failure symptoms and treatment adherence. The score is standardized to a 0- to 100-point range: raw score sum minus lowest possible raw scale score, then divided by the possible range of scores, and finally multiplied by 100. Higher score for each scale indicates better self-maintenance.
Time Frame: Baseline and Six-month follow-up
Population: 6 participants did not complete six months assessment: 4 participants deceased during the study period and 2 participants lost follow-up.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | mHealth
Number analyzed (Participants) | 72
score on a scale
  Baseline | 35 [20 to 47.5]
  Six-month: number analyzed (Participants) | 66
  Six-month | 85 [70 to 85]
Statistical Analysis 1: Comparison: mHealth; Heart failure patients in Uganda were enrolled in an mHealth program at the Uganda Heart Institute. The program intended to promote self-care for heart failure and improve patient healthcare quality of life; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test

2. Primary Outcome: Self-Care for Heart Failure Index, Management
Description: The Self-care of Heart Failure Index (SCHFI) is a measure of self-care defined as a naturalistic decision-making process involving the choice of behaviors that maintain physiological stability (maintenance), the response to symptoms when they occur (management), and confidence in self-care (confidence). The self-care management subscale includes 6 items if patients report any heart failure symptoms in the past month. Then based on the responses on how quick they recognize it as a symptom of heart failure and remedies they tried, the score is standardized to a 0- to 100-point range: raw score sum minus lowest possible raw scale score, then divided by the possible range of scores, and finally multiplied by 100. Higher score for each scale indicates better self-management.
Time Frame: Baseline and Six-month follow-up
Population: The management sub-scale only score if the patient acknowledged having trouble breathing or ankle swelling in the past interval.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | mHealth
Number analyzed (Participants) | 72
score on a scale
  Baseline: number analyzed (Participants) | 52
  Baseline | 20 [10 to 35]
  Six-month: number analyzed (Participants) | 16
  Six-month | 85 [70 to 85]
Statistical Analysis 1: Comparison: mHealth; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test

3. Primary Outcome: Self-Care for Heart Failure Index, Confidence
Description: The Self-care of Heart Failure Index (SCHFI) is a measure of self-care defined as a naturalistic decision-making process involving the choice of behaviors that maintain physiological stability (maintenance), the response to symptoms when they occur (management), and confidence in self-care (confidence). The self-care confidence subscale includes 6 items asking how confident that they can keep themselves free of symptoms, follow treatment advice, recognize changes in their health and etc.. The score is standardized to a 0- to 100-point range: raw score sum minus lowest possible raw scale score, then divided by the possible range of scores, and finally multiplied by 100. Higher score for each scale indicates better self-confidence
Time Frame: Baseline and Six-month follow-up
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | mHealth
Number analyzed (Participants) | 72
score on a scale
  Baseline | 41.2 [23.5 to 52.9]
  Six-month: number analyzed (Participants) | 66
  Six-month | 97.1 [88.2 to 100]
Statistical Analysis 1: Comparison: mHealth; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test

4. Secondary Outcome: EQ-5D-5L, Mobility
Description: Measure Description: Healthcare quality of life will be measured using the 5-level EQ-5D version (EQ-5D-5L). It is a validated instrument appropriate for use in lower and middle income countries. Each of the five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) comprises the EQ-5D descriptive system. We regrouped the 5 levels of perceived problems into binary responses as "no problem" (Level 1), or "Having problems" (Level 2-5).
Time Frame: Baseline and Six-month follow-up visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth
Number analyzed (Participants) | 72
Participants
  Baseline: No Problems | 47
  Baseline: Having Problems | 25
  Six-month: number analyzed (Participants) | 66
  Six-month: No Problems | 54
  Six-month: Having Problems | 12
Statistical Analysis 1: Comparison: mHealth; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.028, Chi-squared; Wilcoxon sign-rank test used to compared baseline outcomes to 6 month outcomes

5. Secondary Outcome: EQ-5D-5L, Self-Care
Description: as for outcome 4
Time Frame: Baseline and Six-month follow-up visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth
Number analyzed (Participants) | 72
Participants
  Baseline: No problems | 42
  Baseline: Having problems | 30
  Six-month: number analyzed (Participants) | 66
  Six-month: No problems | 58
  Six-month: Having problems | 8
Statistical Analysis 1: Comparison: mHealth; Test type: Superiority; p < 0.001, Chi-squared

6. Secondary Outcome: EQ-5D-5L, Usual Activities
Description: as for outcome 4
Time Frame: Baseline and Six-month follow-up visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth
Number analyzed (Participants) | 72
Participants
  Baseline: No problems | 33
  Baseline: Having problems | 39
  Six-month: number analyzed (Participants) | 66
  Six-month: No problems | 54
  Six-month: Having problems | 12
Statistical Analysis 1: Comparison: mHealth; Test type: Superiority; p < 0.001, Chi-squared

7. Secondary Outcome: EQ-5D-5L, Pain or Discomfort
Description: as for outcome 4
Time Frame: Baseline and Six-month follow-up visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth
Number analyzed (Participants) | 72
Participants
  Baseline: No problems | 42
  Baseline: Having problems | 30
  Six-month: number analyzed (Participants) | 66
  Six-month: No problems | 45
  Six-month: Having problems | 21
Statistical Analysis 1: Comparison: mHealth; Test type: Superiority; p = 0.23, Chi-squared

8. Secondary Outcome: EQ-5D-5L, Anxiety or Depression
Description: as for outcome 4
Time Frame: Baseline and Six-month follow-up visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth
Number analyzed (Participants) | 72
Participants
  Baseline: No problems | 44
  Baseline: Having problems | 28
  Six-month: number analyzed (Participants) | 66
  Six-month: No problems | 57
  Six-month: Having problems | 9
Statistical Analysis 1: Comparison: mHealth; Test type: Superiority; p < 0.001, Chi-squared

9. Secondary Outcome: EQ-5D-5L, VAS
Description: The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the 100 indicates 'The best health you can imagine' and 0 means 'The worst health you can imagine'.
Time Frame: Baseline and Six-month follow-up visit
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on the visual analogue scale
Arm/Group | mHealth
Number analyzed (Participants) | 72
score on the visual analogue scale
  Baseline | 70 [50 to 80]
  Six-month: number analyzed (Participants) | 66
  Six-month | 80 [75 to 90]
Statistical Analysis 1: Comparison: mHealth; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test

10. Secondary Outcome: Six-Minute Walk Test, Total Distance
Description: Patients' functional capacity will be assessed using the Six-Minute Walk Test, a widely-used, reproducible exercise test that serves as a strong predictor of morbidity and mortality in heart failure patients. Outcome is measured as a distance in meters. Possible range is 0-700m. Healthy range is considered 400-700m but may not be normative for all populations, including people with chronic diseases. In this study difference in distance (meters) will be examined across visits, with a lower score reflecting worse function.
Time Frame: Baseline and Six-month follow-up visit
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Meters
Arm/Group | mHealth
Number analyzed (Participants) | 72
Meters
  Baseline | 320.3 [220.0 to 360.0]
  Six-month: number analyzed (Participants) | 66
  Six-month | 340.0 [280.0 to 420.0]
Statistical Analysis 1: Comparison: mHealth; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test

11. Secondary Outcome: Left Ventricular Ejection Fraction
Description: Left ventricular ejection fraction (LVEF) is a widely-recognized clinical prognostic marker for heart failure patients. It is measured as a percentage. Possible range is 0-100. Low is <50%. High is >=50%. LVEF is measured by echocardiogram using Simpson biplane formula
Time Frame: Baseline and Six-month follow-up visit
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage of Left Ventricular Ejection
Arm/Group | mHealth
Number analyzed (Participants) | 72
Percentage of Left Ventricular Ejection
  Baseline | 30 [23.5 to 34.5]
  Six-month: number analyzed (Participants) | 66
  Six-month | 33.0 [21.0 to 40.0]
Statistical Analysis 1: Comparison: mHealth; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test

12. Secondary Outcome: Frequency of Acute Care Visits
Description: Patients will be asked to report how often they required acute care for their heart failure outside of their usual care. This outcome is the frequency of acute care visits as categorical variable: 0, 1 and ≥2. Possible range is 0-31.
Time Frame: Baseline and Six-month follow-up visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth
Number analyzed (Participants) | 72
Participants
  Baseline: 0 | 56
  Baseline: 1 | 12
  Baseline: ≥2 | 4
  Six-month: number analyzed (Participants) | 66
  Six-month: 0 | 60
  Six-month: 1 | 6
  Six-month: ≥2 | 0
Statistical Analysis 1: Comparison: mHealth; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | mHealth
All-Cause Mortality (participants affected / at risk) | 4/72
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT04426630/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT04426630/ICF_001.pdf